CLINICAL TRIAL: NCT01825200
Title: Comparison of the Safety of Flublok® Versus Licensed Inactivated Influenza Vaccine in Healthy, Medically Stable Adults ≥ 50 Years of Age
Brief Title: Comparison of the Safety of Flublok® Versus Licensed IIV in Healthy, Medically Stable Adults ≥ 50 Years of Age
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Protein Sciences Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: PSC11
Record Dates: First submitted 2013-03-11; First posted 2013-04-05 (Estimated); Results first posted 2015-02-18 (Estimated); Last update posted 2015-02-18 (Estimated); Status verified 2015-01

CONDITIONS: Influenza
Keywords: Influenza
MeSH Terms: conditions — Influenza, Human | interventions — FluBlok; Afluria

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Flublok (Active Comparator): Flublok containing 3x45µg (135µg total) of recombinant hemagglutinin (rHA) derived from influenza A/H1N1 and A/H3N2 and influenza B viruses in a total volume of 0.5 mL
  Interventions: Biological: Flublok
- Afluria (Placebo Comparator): Afluria, containing 3x15µg (45µg total), of trivalent, inactivated influenza vaccine (licensed IIV) containing influenza antigen derived from A/H1N1 and A/H3N2 and influenza B viruses in a total volume of 0.5 mL
  Interventions: Biological: Afluria

INTERVENTIONS:
Biological: Flublok — A Biologics Licensing Application (BLA) for Flublok was approved by the FDA for influenza immunization of adults 18-49 years of age. Flublok is produced using recombinant technology under serum-free conditions.
  Arms: Flublok
Biological: Afluria — Afluria is approved for use in persons 5 years of age and older and is produced by inactivation and disruption of live influenza virus grown in embryonated chicken eggs.
  Arms: Afluria

SUMMARY:
The hypothesis for this trial is that the incidence of a pre-defined composite of common systemic hypersensitivity adverse events for Flublok recipients is non-inferior to that reported for licensed IIV recipients. Another hypothesis is that the safety and reactogenicity of Flublok is clinically acceptable, i.e. consistent with the overall safety profiles previously observed with Flublok and with the licensed comparator.

DETAILED DESCRIPTION:
The Advisory Committee on Immunization Practices (ACIP) recommends that all people aged 6 months and older be immunized to prevent influenza. Currently the only approved influenza vaccine across the entire age group is inactivated influenza vaccine (IIV). A Biologics Licensing Application (BLA) for Flublok was approved by the FDA for influenza immunization of adults 18-49 years of age. Additional safety and, ultimately efficacy, data is needed to support use in adults ≥50 years of age, an important age group as adults ≥65 years of age are among those at increased risk of influenza complications.

ELIGIBILITY:
Inclusion Criteria:

1. Ambulatory adults aged 50 years and older
2. Medically stable, as determined by medical history and targeted physical examination based on medical history, if appropriate
3. Able to understand and comply with planned study procedures
4. Provides written informed consent prior to initiation of any study procedure.

Exclusion Criteria:

1. Known contraindication to either study vaccine (see product package inserts)
2. Receipt of any other influenza or other vaccine within 30 days prior to enrollment in this study.
3. Receipt of any new medication within 30 days prior to enrollment in this study
4. Plans to participate in any investigation involving an investigational product during this study.
5. Pre-existence of atopic dermatitis or any other cutaneous disorder that could complicate the evaluation of potential primary endpoints.
6. Any clinical or social circumstance that in the opinion of the investigator could interfere with compliance with study procedures or interfere with the interpretation of clinical data.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2640 (Actual)
Dates: Start 2013-03; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brandon Essink, MD, Principal Investigator — Meridian Clinical Research; Paul Bradley, MD, Principal Investigator — Meridian Clinical Research; William Seger, MD, Principal Investigator — Benchmark Research; Darrell Herrington, DO, Principal Investigator — Benchmark Research; George Bauer, MD, Principal Investigator — Benchmark Research; Frank Eder, MD, Principal Investigator — Regional Clinical Research; Treva Tyson, MD, Principal Investigator — Wake Research; Bob Weiss, MD, Principal Investigator — Maine Research Associates, LLC; Jeffrey Rosen, MD, Principal Investigator — Clinical Research of South Florida; Joe Blumenau, MD, Principal Investigator — Research Across America; Steven Folkerth, MD, Principal Investigator — Clinical Research Center of Nevada, LLC; Leah Schmidt, DO, Principal Investigator — Genova Clinical Research; Eric Sheldon, Principal Investigator — Miami Research Associates; Alan C. Wine, MD, Principal Investigator — Rapid Medical Research, Inc.; Terry Poling, MD, Principal Investigator — Heartland Research Associates, LLC
Locations (14):
- United States (14):
  - Genova Clinical Research, Tucson, Arizona
  - Clinical Research of South Florida, Coral Gables, Florida
  - Meridian Clinical Research, Savannah, Georgia
  - Heartland Research Associates, LLC, Wichita, Kansas
  - Benchmark Research, Metairie, Louisiana
  - Maine Research Associates, LLC, Auburn, Maine
  - Meridian Clinical Research, Omaha, Nebraska
  - Clinical Research Center of Nevada, LLC, Las Vegas, Nevada
  - Regional Clinical Research, Binghamton, New York
  - Wake Research, Raleigh, North Carolina
  - Rapid Medical Research, Inc., Cleveland, Ohio
  - Research Across America, Dallas, Texas
  - Benchmark Research, Fort Worth, Texas
  - Benchmark Research, San Angelo, Texas

REFERENCES:
- [Derived] Izikson R, Leffell DJ, Bock SA, Patriarca PA, Post P, Dunkle LM, Cox MM. Randomized comparison of the safety of Flublok((R)) versus licensed inactivated influenza vaccine in healthy, medically stable adults >/= 50 years of age. Vaccine. 2015 Nov 27;33(48):6622-8. doi: 10.1016/j.vaccine.2015.10.097. Epub 2015 Nov 1. PMID 26529070
- See also: Related Info — http://proteinsciences.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited at outpatient medical clinics over a period of five weeks.
Groups:
- Flublok: Flublok containing 3x45µg (135µg total) of rHA0 derived from influenza A/H1N1 and A/H3N2 and influenza B viruses in a total volume of 0.5mL
  Flublok: A Biologics Licensing Application (BLA) for Flublok was approved by the FDA for influenza immunization of adults 18-49 years of age. Flublok is produced using recombinant technology under serum-free conditions.
- Afluria: Afluria, containing 3x15µg (45µg total), of trivalent, inactivated influenza vaccine (licensed IIV) containing influenza antigen derived from A/H1N1 and A/H3N2 and influenza B viruses in a total volume of 0.5mL
  Afluria: Afluria is approved for use in persons 5 years of age and older and is produced by inactivation and disruption of live influenza virus grown in embryonated chicken eggs.
Period: Overall Study
Arm/Group | Flublok | Afluria
Started | 1319 | 1321
Completed | 1314 | 1314
Not Completed | 5 | 7
Not completed — Lost to Follow-up | 5 | 6
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Population: The primary analysis population includes all randomized subjects who received a dose of study vaccine and for whom some safety data were available after administration of vaccine. Subjects were analyzed according to the vaccine received, regardless of whether this was the treatment group to which they were randomized.
Groups:
- Total: Total of all reporting groups
Arm/Group | Flublok | Afluria | Total
Number analyzed (Participants) | 1314 | 1313 | 2627
Age, Continuous [Mean (Full Range); unit: years] | 64 [50 to 99] | 64 [50 to 93] | 64 [50 to 99]
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 672 | 665 | 1337
  >=65 years | 642 | 648 | 1290
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 730 | 725 | 1455
  Male | 584 | 588 | 1172
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 8 | 6 | 14
  Asian | 7 | 5 | 12
  Native Hawaiian or Other Pacific Islander | 1 | 2 | 3
  Black or African American | 197 | 212 | 409
  White | 1098 | 1083 | 2181
  More than one race | 3 | 5 | 8
  Unknown or Not Reported | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 105 | 99 | 204
  Not Hispanic or Latino | 1209 | 1214 | 2423
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 1314 | 1313 | 2627

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Common Hypersensitivity Reactions as Measure of Safety
Description: Number of participants who experience a pre-defined common systemic hypersensitivity adverse event, including rash, urticaria, swelling or edema through Day 30 post-vaccine administration.
Time Frame: 30 Days
Population: The primary analysis population, includes all randomized subjects who received a dose of study vaccine and for whom some safety data were available after administration of vaccine. Subjects were analyzed according to the vaccine received, regardless of whether this was the treatment group to which they were randomized.
Measure: Number; unit: participants
Arm/Group | Flublok | Afluria
Number analyzed (Participants) | 1314 | 1313
participants | 31 | 21

2. Secondary Outcome: Subjects With at Least One Unsolicited Adverse Event in the 30 Days Following Vaccine Administration
Description: Subjects with at least one serious adverse event and subjects with at least one medically-attended unsolicited adverse event occurring during the 30 days following vaccine administration
Time Frame: 30 Days
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Flublok | Afluria
Number analyzed (Participants) | 1314 | 1313
participants
  Serious Adverse Events (SAEs) | 5 | 10
  Medically-Attended Unsolicited Adverse Events | 53 | 51

3. Secondary Outcome: Number of Participants With Local and Systemic Events Reported as a Measure of Safety
Description: Number of solicited local and systemic events of reactogenicity reported with the help of a memory aid during the seven days following vaccine administration.
Time Frame: 7 Days
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Flublok | Afluria
Number analyzed (Participants) | 1314 | 1313
participants | 432 | 480

4. Secondary Outcome: Subjects With at Least One Hypersensitivity Event Reported on Day 0 and Days 0-7 Following Vaccine Administration as a Measure of Safety
Description: Subjects with at least one pre-defined common systemic hypersensitivity adverse event, including rash, urticaria, swelling or non-dependent edema on Day 0 and for Days 0 to 7 following vaccine administration
Time Frame: 7 Days
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Flublok | Afluria
Number analyzed (Participants) | 1314 | 1313
participants
  Day 0 | 5 | 3
  Days 0-7 | 25 | 12

ADVERSE EVENTS:
Time Frame: 30 days following vaccine administration
Description: Adverse Events were reviewed by Investigators and by the Medical Monitor. Assessments of causality were conducted by both reviewers.
Arm/Group | Flublok | Afluria
Serious Adverse Events (participants affected / at risk) | 5/1314 | 10/1313
Other Adverse Events (participants affected / at risk) | 20/1314 | 16/1313
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Flublok (N=1314) | Afluria (N=1313)
Cerebellar Stroke Syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 2 (2)
Myocardial Infarction (Cardiac disorders) | 1 (1) | 2 (2)
Diabetic Ketoacidosis (Endocrine disorders) | 0 (0) | 1 (1)
Alcoholic Hepatitis (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Leg Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Salivary Gland Tumor (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Hypertension (Cardiac disorders) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Flublok (N=1314) | Afluria (N=1313)
Headache (Nervous system disorders) | 8 (8) | 12 (12)
Diarrhea (Gastrointestinal disorders) | 12 (12) | 4 (4)

LIMITATIONS AND CAVEATS:
Rash, urticaria, swelling and edema were self-reported by subjects and most were not observed by investigators. Review by independent experts indicated that 42 of 52 subject-reported events did not represent Type 1 (IgE-mediated) hypersensitivity.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less